CLINICAL TRIAL: NCT01598610
Title: Performance of the CONTOUR® PLUS Blood Glucose Monitoring System With CONTOUR® PLUS Strip
Brief Title: Performance Evaluation of an Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2012-002-01
Record Dates: First submitted 2012-05-13; First posted 2012-05-15 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Untrained subjects with diabetes use CONTOUR® PLUS Investigational BG Monitoring System.
  Interventions: Device: CONTOUR® PLUS Investigational BG Monitoring System

INTERVENTIONS:
Device: CONTOUR® PLUS Investigational BG Monitoring System — Untrained subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the CONTOUR® PLUS Investigational BG Monitoring System. Study staff test subject venous blood. All Blood Glucose (BG) results are compared to a reference laboratory glucose method.

SUMMARY:
The purpose of this study is to demonstrate that untrained subjects who have diabetes can operate the Investigational Blood Glucose Monitoring System (BGMS) and obtain valid glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* Type 1 or type 2 diabetes
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Pregnancy
* Hemophilia or any other bleeding disorder
* Previously participated in a study using the CONTOUR PLUS system
* Working for a medical laboratory, hospital or other clinical setting that involves training on and clinical use of blood glucose monitors.
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company.
* A condition, which in the opinion of the investigator, would put the person or study conduct at risk (reason for exclusion will be clearly documented by investigator or designee).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip D Toth, MD, FACP, Principal Investigator — Midwest Institute For Clinical Research; Michael Caswell, PhD, Principal Investigator — Consumer Product Testing Co.
Locations (2):
- United States (2):
  - Midwest Institute For Clinical Research, Indianapolis, Indiana
  - Consumer Product Testing Co., Fairfield, New Jersey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 220
Completed | 219
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 220
Age, Continuous [Mean (Full Range); unit: years] | 60 [26 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 102
Region of Enrollment [Number; unit: participants]
  United States | 220

OUTCOME MEASURES:

1. Primary Outcome: Percent of Self-Test Fingerstick Blood Glucose Results Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. BG results are used to calculate the number of BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma) of the reference method results.
Time Frame: 1 hour
Population: 216 (220-4) blood test results were analyzed. Blood data for 2 subjects were not evaluable because time, defined in protocol, was exceeded between meter test and blood sample preparation for reference method. No fingerstick results were obtained for 2 subjects.
Measure: Number; unit: percentage of BG Test Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 216
percentage of BG Test Results | 100

2. Secondary Outcome: Percent of Glucose Results From Alternative Site Testing (AST) of the Palm Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test Alternative Site (AST) Palm blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS AST results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. BG results are used to calculate the number of AST BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma) of the reference method results.
Time Frame: 1 hour
Population: 213 (220-7) blood test results were analyzed. Four(4) subjects had low blood sugar and AST results were not evaluable per protocol. One(1) subject with low blood sugar (AE) did not attempt AST testing per protocol. No AST palm results were obtained for 2 subjects.
Measure: Number; unit: percentage of BG Test Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 213
percentage of BG Test Results | 98.1

3. Secondary Outcome: Percent of Venous Blood Glucose Results Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method
Description: Study staff tested subject venous blood using an investigational Blood Glucose Monitoring System (BGMS). Venous BGMS results are compared with venous plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. Venous plasma BG results are used to calculate the number of BGMS results within +/- 15mg/dL (<75mg/dL YSI venous plasma) or +/- 20% (>=75mg/dL YSI venous plasma) of the reference method results.
Time Frame: 1 hour
Population: 213 (220-7) blood test results were analyzed. Venipuncture was unsuccessful for 6 subjects. Blood data for 1 subject was not evaluable because time, defined in protocol, was exceeded between meter test and blood sample preparation for reference method.
Measure: Number; unit: percentage of BG Test Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 213
percentage of BG Test Results | 99.5

4. Secondary Outcome: Percent of Self-Test Fingerstick Blood Glucose Results Within +/- 5to15mg/dL (<100mg/dL) or Within +/- 5to15% (>=100mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. BG results are used to calculate the number of BGMS results within +/- 5to15mg/dL (<100mg/dL YSI capillary plasma) or +/- 5to15% (>=100mg/dL YSI capillary plasma) of the reference method results.
Time Frame: 1 hour
Population: 108 (110-2) blood test results from one test strip lot were analyzed. Blood data for 1 subject was not evaluable because time, defined in protocol, was exceeded between meter test and blood sample preparation for reference method. No fingerstick result was obtained for 1 subject.
Measure: Number; unit: percentage of BG Test Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 108
percentage of BG Test Results
  % within +/-15mg/dL(<100mg/dL) or 15% (>=100mg/dL) | 98.2
  w/in +/-12.5mg/dL(<100mg/dL) or 12.5% (>=100mg/dL) | 93.5
  w/in +/-10mg/dL(<100mg/dL) or +/- 10% (>=100mg/dL) | 86.1
  w/in +/-5mg/dL(<100mg/dL) or +/- 5% (>=100mg/dL) | 53.7

5. Secondary Outcome: Percent of Subject Fingerstick BG Results Within +/- 15mg/dL (<75mg/dL) or Within +/- 20% (>=75mg/dL) of Laboratory Glucose Method When Tested by Study Staff
Description: Study staff test subject fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. BG results are used to calculate the number of BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma) of the reference method results.
Time Frame: 1 hour
Population: 217 (220-3) blood test results were analyzed. Blood data for 2 subjects were not evaluable because time, defined in protocol, was exceeded between meter test and blood sample preparation for reference method. No fingerstick results were obtained for 1 subject.
Measure: Number; unit: percentage of BG Test Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 217
percentage of BG Test Results | 99.5

6. Secondary Outcome: Number of Subject Responses 'Strongly Agree' 'Agree' or 'Neutral' With Questionnaire Statements
Description: Subjects respond to statements read by study staff to provide feedback on the labeling materials and system ease of use. Subjects may respond 'Strongly Agree' 'Agree' 'Neutral' 'Disagree' or 'Strongly Disagree'.
Time Frame: 1 hour
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 220
participants
  I found it easy to do a blood test with this meter | 215
  Meter display(test result) is easy to see and read | 220
  It was easy to understand my test results. | 218
  I like the overall meter design. | 218
  I find the meter easy to handle. | 218
  Easy to handle the individual test strips. | 218
  Instructions (User Guide) easy to understand. | 218
  Instructions clearly explain how to run a test. | 220
  Instructions clearly explain meter error messages. | 218

ADVERSE EVENTS:
Arm/Group | Intended Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/220
Other Adverse Events (participants affected / at risk) | 2/220
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the Monitoring System (N=220)
hypoglycemia (Endocrine disorders) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days